CLINICAL TRIAL: NCT05499533
Title: Hybrid Funnel Technique vs Conventional Drill Osteotomy, a Novel Approach for Implant Site Preparation
Brief Title: Hybrid Funnel Technique a Innovative Technique for Implant Site Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luigi Canullo (Other)
Responsible Party: Sponsor-Investigator, Luigi Canullo, principal investigator, Studio Odontoiatrico Associato Dr. P. Cicchese e L. Canullo
Organization: Studio Odontoiatrico Associato Dr. P. Cicchese e L. Canullo (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABT3
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Missing Teeth; Edentulous Alveolar Ridge; Tooth Loss
Keywords: osteotomy; dental implant; marginal bone loss; implant stability; osteotome; implant site preparation
MeSH Terms: conditions — Anodontia; Tooth Loss | interventions — Osteotomy

STUDY DESIGN:
Intervention Model Description: Once selected, patients will be assigned to one of two treatment groups. (test group- hybrid funnel technique; control group- conventional drill technique) Patients are placed in one of the two treatment groups according to the chronological order in which they will be recruited. Age, sex, surgical implant site (upper, lower, anterior, posterior) and clinical l characteristics will be taken into account to obtain two homogeneous study groups.
  First Hybrid Funnel Technique will be performed, then Conventional drill Technique will be performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid Funnel Technique (Experimental): Hybrid funnel technique for implant site preparation
  Interventions: Procedure: implant site preparation
- Conventional Technique (Active Comparator): Conventional subtractive Drill technique for implant site preparation
  Interventions: Procedure: implant site preparation

INTERVENTIONS:
Procedure: implant site preparation — a hole were created in the edentulous ridge area before implant placement
  Other Names: osteotomy

SUMMARY:
Hybrid Funnel Technique arises from the union of subtractive and non-subtractive techniques for implant site preparation. Hybrid funnel technique is performed with specially designed drills and osteotome. the aim of the study is to examine marginal bone level and implant stability of implants inserted with two different techniques for the surgical implant site preparation.

DETAILED DESCRIPTION:
Overtime several osteotomy techniques were described in literature for surgical implant site preparation and there is a clear dichotomy between expansive and ablative techniques.

The ablative techniques imply the preparation of the implant socket by removing bone: drill osteotomy and ultrasonic osteotomy. Expansive technique for osteotomy has recently been proposed: the osseodensification. Osseodensification, a non-subtractive instrumentation method, involves the use of specific drills or manual osteotomes which determine an expansion of the implant site without bone removal and bone fragments compaction on the walls of implant socket.The aim of the present study is to propose a new approach for the implant site preparation that combines ablative and expansive techniques. The technique proposed is called hybrid funnel techniqueAlthough a variety of techniques are available for implant site preparation, the hypothesis is that Hybrid Funnel technique will be positively adopted to perform osteotomy, exploiting the cancellous bone elastic properties to stabilize the implant and avoiding to stress the cortical area. Primary objectives are to compare hybrid funnel technique and traditional technique on different bone densities and to examine Marginal Bone Level torque insertion value and Implant stability.

ELIGIBILITY:
Inclusion Criteria:

1. Patient needing for post-extraction implant supported restoration in the mandibular or maxillary area
2. ASA 1 E ASA 2
3. Subject is 30-85 years old
4. Patients with healthy periodontal conditions (Treated periodontitis, PI<25%, BoP<25%)
5. Patients that are willing to sign an informed consent and participate in a clinical study

Exclusion Criteria:

1. Absence Type 1-2 post extraction sites
2. Patient ASA 3 or 4
3. Any sites where an implant already failed sites
4. Untreated Periodontitis
5. Allergy declared to one or more medicaments to be used during treatment
6. Pregnancy (confirmed by verbal inquiry)

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Marginal bone loss | 6 months after implant placement
  Radiographic evaluation of the marignal bone level around the implant using a periapical x ray. marginal bone loss is in millimeters and indicates how many millimeters of bone has been lost
Marginal bone loss | 12 months after implant placement
  Radiographic evaluation of the marignal bone level around the implant using a periapical x ray. marginal bone loss is in millimeters and indicates how many millimeters of bone has been lost
Implant stability | immediately after implant placement
  check implant stability using resonant frequency analysis (RFA)
Implant stability | 2 months after implant placement
  check implant stability using resonant frequency analysis (RFA)
Insertion torque curve | During implant placement (T0 baseline)
  The Insertion torque data were recorded and exported as a curve The torque curve records the amount of energy that was needed for arrive at the positioning of the implantunit of measurement of torque is Newton centimeter (Ncm)

CONTACTS AND LOCATIONS:
Locations (1):
- Studio Odont.Associato Dr.P.Cicchese E L.Canullo, Rome, Italy/Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yeo IL. Modifications of Dental Implant Surfaces at the Micro- and Nano-Level for Enhanced Osseointegration. Materials (Basel). 2019 Dec 23;13(1):89. doi: 10.3390/ma13010089. PMID 31878016
- [Background] Trisi P, Berardini M, Falco A, Podaliri Vulpiani M. New Osseodensification Implant Site Preparation Method to Increase Bone Density in Low-Density Bone: In Vivo Evaluation in Sheep. Implant Dent. 2016 Feb;25(1):24-31. doi: 10.1097/ID.0000000000000358. PMID 26584202
- [Background] Toia M, Stocchero M, Cecchinato F, Corra E, Jimbo R, Cecchinato D. Clinical Considerations of Adapted Drilling Protocol by Bone Quality Perception. Int J Oral Maxillofac Implants. 2017 Nov/Dec;32(6):1288-1295. doi: 10.11607/jomi.5881. PMID 29140373
- [Background] Stacchi C, Vercellotti T, Torelli L, Furlan F, Di Lenarda R. Changes in implant stability using different site preparation techniques: twist drills versus piezosurgery. A single-blinded, randomized, controlled clinical trial. Clin Implant Dent Relat Res. 2013 Apr;15(2):188-97. doi: 10.1111/j.1708-8208.2011.00341.x. Epub 2011 Apr 19. PMID 21682844
- [Background] Ivanova V, Chenchev I, Zlatev S, Mijiritsky E. Correlation between Primary, Secondary Stability, Bone Density, Percentage of Vital Bone Formation and Implant Size. Int J Environ Res Public Health. 2021 Jun 30;18(13):6994. doi: 10.3390/ijerph18136994. PMID 34208849
- [Background] Alifarag AM, Lopez CD, Neiva RF, Tovar N, Witek L, Coelho PG. Atemporal osseointegration: Early biomechanical stability through osseodensification. J Orthop Res. 2018 Sep;36(9):2516-2523. doi: 10.1002/jor.23893. Epub 2018 Mar 30. PMID 29537128